CLINICAL TRIAL: NCT05895370
Title: A Phase 1 Study to Assess the Feasibility and Safety of Tumor HPV-E6/E7-Targeting T Cell Suspension for Intravenous Infusion (HPV-T) in Patients With HPV-16 Positive Recurrent or Metastatic Solid Tumor
Brief Title: HPV-T in HPV-16 Positive Recurrent or Metastatic Solid Tumors
Acronym: GI-HPVT-01
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: BGI, China (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGI-005
Record Dates: First submitted 2023-05-31; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Solid Tumor
Keywords: HPV-16 Positive; Adoptive T Cell Therapy; Recurrent or Metastatic Cervical Cancer; HPV-T
MeSH Terms: conditions — Recurrence; Uterine Cervical Neoplasms | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPV-T (Experimental): Participants in the 2 dose groups will receive HPV-T injections of 5×10^9 and 1.5×10^10 cells intravenously each time.
  Interventions: Biological: HPV-T; Drug: Interleukin-2

INTERVENTIONS:
Biological: HPV-T — Participant will receive HPV-T iv on day 0. One time of cell infusion constitute a cycle, each participant receives up to four cycles of treatment
Drug: Interleukin-2 — 500,000IU/m^2 SC, after each cell infusion, IL-2 will start within 24 hours and every 8-12 hours for up to 6 doses.
  Other Names: IL-2

SUMMARY:
The purpose of this protocol is to evaluate the feasibility and safety of HPV-T in HPV 16 positive recurrent or metastatic solid tumor patients.

DETAILED DESCRIPTION:
In this study, HPV-T cells will be cultured from mononuclear cells collected from participant's peripheral blood in the laboratory and they will be given back to the participant intravenously. The use of HPV-T cells involves a combination of IL-2, which is a drug used to help the body's response to treatment on the immune system. A medium dose regimen of IL-2 will be given after the participant receives the infusion of the T-cells.

Each HPV-T cell reinfusion is a treatment cycle, and each participant will receive a maximum of four cycles of HPV-T treatment. Whether the participant receives the next cycle of treatment depends on the efficacy of the previous HPV-T treatment, which is assessed by imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than or equal to 18 years of age and less than or equal to 75 years of age; all genders.
2. Confirmed diagnosis of recurrent of metastatic solid tumor and at least one measurable lesion.
3. HLA type is HLA-A0201.
4. HPV 16 positive.
5. Patients who failed or were intolerant to standard first-line treatment.
6. Possess venous access for mononuclear cell collection or intravenous blood collection.
7. Clinical performance status of ECOG is 0 or 1.
8. Possess venous access for mononuclear cell collection or intravenous blood collection.
9. Patients who are able to cooperate to observe adverse reactions and the effect of the treatment,expected lifetime is greater than six month.
10. Patients of both genders must be willing to practice birth control from the time of enrollment to three months after treatment on this study,a fertile woman must have a negative pregnancy test.
11. The laboratory test values and the functions of important organs meet the following requirements:

1#Serology: HIV antibody(-), hepatitis B DNA(-), hepatitis C antibody(-) and no active syphilis infection; 2#Hematology: Absolute neutrophil count is greater than or equal to 1.5×10^9/L; WBC is greater than or equal to 3×10^9/L; lymphocyte count is greater than or equal to 0.8×10^9/L; Platelet count is greater than or equal to 100×10^9/L; Hemoglobin is greater than or equal to 85g/L ; 3#Chemistry: Serum ALT/AST is less than or equal to 3 times ULN,except in patients with liver metastasis who must have ALT/AST less than or equal to 5 times ULN; Serum Creatinine is less than or equal to 1.5 times ULN ; Total bilirubin is less than or equal to 1.5 times ULN, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3 times ULN; 4#Blood Clotting Parameters:Prothrombin Time(PT) and International Normalised Ratio (INR) are less than or equal to 1.5 times ULN;Activated Partial Thromboplastin Time (APTT) is less than or equal to 1.5 times ULN;For subjects who frequently take anticoagulant drugs,their blood clotting parameters can meet the value range adoptive to this special population; 5#Left ventricular ejection fraction#LVEF#is more than or equal to 50%. 12. More than four weeks must have elapsed since any prior systemic therapy (except for bridging therapy) at the time the patient receives the lymphodepletion regimen, and toxicities must have recovered to grade 1 or less (except for toxicities such as alopecia or vitiligo)

Exclusion Criteria:

1. Pregnant or lactating women.
2. History of severe immediate hypersensitivity reaction to HPV-T and any of the agents used in this study.
3. Participants with a history of organ transplantation.
4. Participants with brain metastases.
5. Any active autoimmune disease or participants with a history of autoimmune diseases that have been assessed by the investigator to be unsuitable for this study. Including but not limited to the following diseases: such as systemic lupus erythematosus, immune related neuropathy, multiple sclerosis, Guillain Barre syndrome, myasthenia gravis, connective tissue diseases, inflammatory bowel diseases(Crohn's disease and ulcerative colitis), excluding vitiligo, eczema, type I diabetes, rheumatoid arthritis and other joint diseases, Sjogren's syndrome and controlled psoriasis by local medication.
6. Active systemic infections, for example, acute infections requiring systemic antibiotic, antiviral, or antifungal treatment occur within 2 weeks before enrollment.
7. Severe liver and kidney function damage(given treatment is still uncontrollable, and biochemical indicators cannot meet the Exclusion Criteria of 11th), uncontrollable diabetes, pulmonary fibrosis, interstitial lung disease, acute lung disease, or poorly controlled hypertension (systolic pressure>160mmHg and/or diastolic pressure>90mmHg); active cardiovascular and cerebrovascular diseases, such as acute stroke, myocardial infarction, unstable angina, congestive heart failure rated as Grade II or above by the New York Heart Association, severe cardiac arrhythmias that cannot be controlled with medication, electrocardiograms show significant abnormalities (three consecutive times with an interval of at least 5 minutes) which have been assessed by the investigator that affect subsequent cellular treatment; mental illness and drug abuse, or any situation that the investigator assessments may increase the risk of this study.
8. Participants plan to receive glucocorticoid (the dose of prednisone or alternative drug is more than 10mg per day) or other immunosuppressant within 4 weeks before the administration of lymphocyte clearance. Tips: when there is no active autoimmune disease, it is allowed to use prednisone or alternative drug with a dose less than 10 mg per day; Allowing participants to use topical, ocular, intra articular, intranasal, and inhaled glucocorticoids for treatment.
9. Participants plan to receive immunomodulatory drugs (such as interferon, GM-CSF, thymosin, gamma globulin, excluding IL-2) within 4 weeks before the administration of lymphocyte clearance.
10. The investigator assessed that the subject was unable or unwilling to comply with the requirements of the study protocol.
11. With a history of other malignant tumors.
12. The participant has any disease or medical condition that may affect the safety or effectiveness evaluation of the study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2024-12-13 (Estimated); Study Completion 2025-04-13 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as assessed by CTCAE v5.0 | Up to 24 months
  Toxicity will be assessed within 4 weeks of the HPV-T transfer.

SECONDARY OUTCOMES:
Number of Participants With Objective Response | Up to 24 months
  Participants displaying objective response associated with the treatment regimen per Response Evaluation Criteria in Solid Tumors (RECIST v.1.1). The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria. Disease control rate (DCR), Duration of Response (DOR), Overall Survival(OS) and Progression-free survival (PFS) will be also evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China